CLINICAL TRIAL: NCT03898973
Title: Response to Inactivated Influenza Vaccine in Lymph Tissue and Blood
Acronym: FLU-LN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Were not able to enroll participants
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 50328
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2022-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Phase (Other): Participants will be given the current year's a quadrivalent inactivated influenza vaccine (IIV)
  Interventions: Biological: Quadrivalent inactivated influenza vaccine (IIV)

INTERVENTIONS:
Biological: Quadrivalent inactivated influenza vaccine (IIV) — Intramuscular Injection. Participants will receive the inactivated flu vaccine into anterior quadriceps.
  Other Names: Fluzone Quadrivalent

SUMMARY:
This is one project of a larger ongoing study related to the immune system's response to the flu virus. This study is designed to determine how immune memory develops at the actual site of exposure, and how immunization may alter this process.

DETAILED DESCRIPTION:
This is a Phase IV study of licensed influenza vaccines with up to 50 volunteers, 20-75 years of age.

Each volunteer will participate for approximately 1 week including enrollment, vaccination, and completion of sample collection.

The study has a total of 3 visits.

Study Procedures:

Screening Visit: Procedures during this visit are: Informed consent process, assess eligibility collect relevant clinical data and obtain 10 mL of blood to ensure the FNA will be safe (acceptable CBC and PT/PTT).

Visit 1: Vaccination Visit:

Eligible subjects will return and have a 20 mL blood sample. Participants will receive the inactivated flu vaccine into the right anterior quadriceps. Volunteers will be monitored for at least 15 minutes after study vaccination.

Visit 2: FNA Procedure: Seven days after vaccination the participant will return for another collection of 20 ml of blood and a fine needle aspiration of a right inguinal lymph node under ultrasound guidance by a trained pathologist.

ELIGIBILITY:
Inclusion Criteria:

1. 20-75-year-old male and female patients
2. Body mass index (BMI) 20-35 kg/m2
3. Acceptable laboratory values: Absolute neutrophil count (ANC) > 750 cells/mm3; Hemoglobin >10 g/dL; Platelet count >75,000/mm3; Partial thromboplastin time (PTT) >1.2x ULN; Prothrombin time (PT) >1.2x ULN
4. Willing and able to complete the informed consent process
5. Availability for follow-up for the planned duration of the study
6. Acceptable medical history by review of inclusion/exclusion criteria

Exclusion Criteria:

1. Prior off-study vaccination with seasonal influenza vaccine within three months of study vaccination
2. Life-threatening reactions to previous influenza vaccinations
3. Allergy to egg or egg products or to vaccine components
4. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
5. History of immunodeficiency (including HIV infection)
6. Known or suspected impairment of immunologic function; may include significant liver disease, diabetes mellitus treated with insulin or moderate to severe renal disease
7. Chronic Hepatitis B or C.
8. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
9. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
10. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator might jeopardize volunteer safety or compliance with the protocol.
11. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
12. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg per day), Plavix, or Aggrenox will be reviewed by investigators to determine if study participation would affect the volunteer's safety or compliance with the protocol.
13. Receipt of blood or blood products within the past 6 months or planned used during the study.
14. A medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
15. Receipt of an inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last annual study visit (~ 28 days after study vaccination)
16. Receipt of a live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 28 days after study enrollment)
17. Need for allergy immunization (that cannot be postponed) until after the last study visit.
18. History of Guillain-Barre# syndrome
19. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
20. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or donation of platelets within 2 weeks of enrollment or planned donation prior to completion of the last visit.
21. Pregnancy
22. Any condition which, in the opinion of the investigator, might interfere with volunteer safety,

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
HAI titer | Day 7 after vaccination
  This measures response to influenza vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Lane building L134, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No